## Statistical Analysis Plan Cover Page

A Pilot Study to Assess <u>WATCHMAN FLX<sup>TM</sup></u> Implants by Cardiac <u>C</u>omputed <u>T</u>omography, Magnetic Resonance Imaging and Transesophageal Echocardiography: WATCHMAN FLX<sup>TM</sup> CT

## WATCHMAN FLX<sup>TM</sup> CT S2423 CLINICAL INVESTIGATION PLAN

National Clinical Trial (NCT) Identifier Number: NCT05324371

## CONFIDENTIAL DO NOT COPY OR DISTRIBUTE WITHOUT WRITTEN PERMISSION

**Revision History** 

| Revision Number | Notes | Date |
|-----------------|---------------|-------------|
| A | First version | 27-Oct-2022 |